CLINICAL TRIAL: NCT01161511
Title: A Phase 1 Study of XmAb®5574 to Evaluate the Safety, Tolerability, and Pharmacokinetics in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Safety and Tolerability of XmAb®5574 in Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb5574-01
Record Dates: First submitted 2010-07-08; First posted 2010-07-13 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL; CD19
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tafasitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): XmAb5574
  Interventions: Biological: XmAb5574

INTERVENTIONS:
Biological: XmAb5574 — Intravenous infusion of XmAb5574 administered weekly during two 28-day cycles with an additional dose being administered during the first week of Cycle 1. (Cycle 1 on Days 1, 4, 8, 15, 22; Cycle 2 on Days 1, 8, 15, 22)

SUMMARY:
This is an open-label, multi-dose, single-arm, Phase 1, dose-escalation study of XmAb5574. The study was conducted to identify the maximum tolerated dose (MTD) and/or recommended dose(s) (RD) for further study, to characterize safety and tolerability, to characterize PK, PD and immunogenicity, and to evaluate preliminary antitumor activity of XmAb5574 in patients with relapsed or refractory CLL/SLL.

ELIGIBILITY:
Inclusion Criteria:

* relapsed or refractory CLL/SLL
* at least 18 years of age
* able to receive outpatient treatment and follow-up at the treating institution
* completed all CLL therapies > 4 weeks prior to first study dose

Exclusion Criteria:

* previously treated with an anti-CD19 antibody therapy
* undergone prior allogeneic stem cell transplantation within 6 months or having active graft versus host disease
* active Richter's syndrome
* designated Class III or IV by the New York Heart Association (NYHA) criteria
* history of myocardial infarction or stroke within the last 6 months
* active viral, bacterial, or systemic fungal infection requiring treatment
* HIV or Hepatitis C positive
* Hepatitis B infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicities | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John C Byrd, MD, Principal Investigator — Ohio State University, Columbus, Ohio; Farrukh Awan, MD, Principal Investigator — Georgia Health Sciences University, Augusta, Georgia; Ian W Flinn, MD, PhD, Principal Investigator — Sarah Cannon Research Institute, Nashville, Tennessee
Locations (3):
- United States (3):
  - Medical College of Georgia, Augusta, Georgia
  - The Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- [Derived] Woyach JA, Awan F, Flinn IW, Berdeja JG, Wiley E, Mansoor S, Huang Y, Lozanski G, Foster PA, Byrd JC. A phase 1 trial of the Fc-engineered CD19 antibody XmAb5574 (MOR00208) demonstrates safety and preliminary efficacy in relapsed CLL. Blood. 2014 Dec 4;124(24):3553-60. doi: 10.1182/blood-2014-08-593269. Epub 2014 Oct 9. PMID 25301708